CLINICAL TRIAL: NCT01136369
Title: Clinical Evaluation of LS-03M/LS-04R for the Detection of Sentinel Lymph Node Metastasis From Breast Cancer
Brief Title: Clinical Evaluation of OSNA Breast Cancer System to Test Sentinel Lymph Nodes From Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Sysmex America, Inc. (Industry)
Responsible Party: Carrie Pineda, Sysmex America, Inc
Other Study IDs: OSNA-BC-001
Record Dates: First submitted 2010-06-01; First posted 2010-06-03 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Breast Neoplasms; Breast Diseases
Keywords: metastasis; molecular pathology
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of the tissue homogenate will be retained and may be used for for further testing.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- OSNA Breast Cancer System
  Interventions: Device: OSNA Breast Cancer System

INTERVENTIONS:
Device: OSNA Breast Cancer System — For in vitro diagnostic use only.
  The OSNA Breast Cancer System is an automated semi-quantitative, in vitro diagnostic test for the rapid detection of greater than (>) 0.2 mm metastases in nodal tissue removed from sentinel lymph node biopsies of breast cancer patients. Results from the assay can be used to guide the intra-operative or post-operative decision to remove additional lymph nodes and to aid in patient staging. An assay positive + or ++ result indicates the presence of metastasis (> 0.2 mm). An assay positive ++ result predicts the presence of macrometastasis (> 2 mm).
  Post-operative histological evaluation of permanent sections of the tissue specimen, in accordance with usual diagnostic practice and using the Sysmex lymph node cutting scheme, is required.

SUMMARY:
The study will determine the sensitivity, specificity, negative predictive value and positive predictive value of the OSNA Breast Cancer System by comparing its performance to permanent section Hematoxylin and Eosin (H&E) and IHC staining.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients, over the age of 18, diagnosed pre-surgically with T1 or T2 breast cancer and scheduled for surgery including sentinel node dissection.
* Patients who have read and understand the informed consent form and are capable and willing to provide written informed consent.

Exclusion Criteria:

* Patients diagnosed pre-surgically with large or locally advanced (T3 and T4) breast cancers.
* Patients diagnosed with inflammatory breast cancer.
* Patients diagnosed with ductal carcinoma in situ (DCIS) when breast conserving is to be done.
* Patients who are pregnant, as confirmed by a patient/treating physician interview.
* Patients with suspicious palpable axillary lymph nodes.
* Patients currently being treated for or previously diagnosed with, another type of carcinoma.
* Patients who have undergone prior non-oncologic breast surgery or axillary surgery.
* Patients who have received pre-operative systemic therapy.
* Patients who are incapable of providing written informed consent.
* Patients who have been judged to be inappropriate by a medical care provider (i.e. surgeon, oncologist, pathologists, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a previous diagnosis of breast cancer scheduled for sentinel lymph node dissection.
Sampling Method: Probability Sample
Enrollment: 496 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The study will determine the sensitivity, specificity, negative predictive value and positive predictive value of the OSNA Breast Cancer System by comparing its performance to permanent section staining. | 2 years
The time required to perform the trial method will be measured and evaluated for intra-operative use. | 2 Years

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - John Wayne Cancer Institute, Santa Monica, California
  - WellStar Health Systems, Marietta, Georgia
  - Washington University Medical School, St Louis, Missouri
  - Beth Israel Medical Center, New York, New York
  - Central Carolina Surgery, PA, Greensboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Breast Care Specialist, Inc., Westerville, Ohio
  - Breast Care Specialist, PC, Allentown, Pennsylvania
  - Nashville Breast Center, PC, Nashville, Tennessee
  - Dallas Surgical Group, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas